CLINICAL TRIAL: NCT01374607
Title: Assessment of Highly Sensible T Troponin (Hs-TnT) Assay Compared to Standard Troponin Assay in the Early Detection of Cardiac Ischemia in Patients With Acute Coronary Syndrome
Brief Title: Comparison Between High-sensitivity Cardiac Troponin T and Standard Tnl Assays in Early Cardiac Ischemia Detection
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Chief Nuclear medicine Department, University of Lausanne Hospitals
Other Study IDs: 18/11
Record Dates: First submitted 2011-06-08; First posted 2011-06-16 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; myocardial ischemia; high-sensitivity cardiac troponin T
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is crucial to rapidly identify cardiac ischemia in the care of patients with suspected acute coronary syndrome (ACS). Cardiac troponins are a major factor in the diagnostic of myocardial infarction. New methods have been developed to improve the accuracy of the assay and determine low troponin concentrations. Elecsys® (highly sensible T troponin) TnT-HS assay is supposed to help early detection of myocardial infarction after onset of symptoms. It should therefore shorten the transit time to emergencies by a more rapid intervention or a faster return home. The aim of the study is to compare TnT-HS assay to the standard troponin assay in the detection of early cardiac ischemia in patients with ACS.

DETAILED DESCRIPTION:
Patients with suspected ACS with 2/2 negative results of conventional troponin I assay and 1/3 positive result of highly sensitive troponin assay will have a non invasive cardiac Rb82 PET/CT performed within 24 hours of admission. This exam is recognized by Associations of cardiology for its high sensibility and specificity in coronary disease detection.

ELIGIBILITY:
Inclusion Criteria:

* chest pain of ≥ 5 minutes during the last 24 hours, or other symptoms suggestive of ACS (unstable angina or NSTEMI) with 2 negative standard troponin values(<0.09 µg/L)
* age ≥ 18

Exclusion Criteria:

* patients with ST- segment elevation myocardial infarction (STEMI)
* detection of TnI standard values > 0.09 (limit of positivity) in one of two blood samples (T0 and T6)
* detection of heart disease or extra-cardiac disease that could explain the elevated conventional troponin values
* presence of major organ dysfunction, infection or major underlying medical condition that could compromise the patient's ability to perform a stress test for myocardial ischemia
* cancer with prognosis < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency with chest pain suspect of acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
patients presenting to the emergency for chest pain suspect for ACS currently have 2 troponin assays (Tn I) performed at T0 and T6. The additional value of a high sensitivity cardiac troponin T (Hs-TnT) dosage performed at T0 will be analyzed. | T0 (admission)
patients presenting to the emergency for chest pain suspect for ACS currently have 2 troponin assays (Tn I) performed at T0 and T6. The additional value of a high sensitivity cardiac troponin T (Hs-TnT) dosage performed at T2 will be analyzed. | T2 (2 hours after admission)
patients presenting to the emergency for chest pain suspect for ACS currently have 2 troponin assays (Tn I) performed at T0 and T6. The additional value of a high sensitivity cardiac troponin T (Hs-TnT) dosage performed at T6 will be analyzed. | T6 (6 hours after admission)

SECONDARY OUTCOMES:
major cardiovascular events | at 30 days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Muller, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reichlin T, Hochholzer W, Bassetti S, Steuer S, Stelzig C, Hartwiger S, Biedert S, Schaub N, Buerge C, Potocki M, Noveanu M, Breidthardt T, Twerenbold R, Winkler K, Bingisser R, Mueller C. Early diagnosis of myocardial infarction with sensitive cardiac troponin assays. N Engl J Med. 2009 Aug 27;361(9):858-67. doi: 10.1056/NEJMoa0900428. PMID 19710484
- [Derived] Morawiec B, Fournier S, Tapponnier M, Prior JO, Monney P, Dunet V, Lauriers N, Recordon F, Trana C, Iglesias JF, Kawecki D, Boulat O, Bardy D, Lamsidri S, Eeckhout E, Hugli O, Muller O. Performance of highly sensitive cardiac troponin T assay to detect ischaemia at PET-CT in low-risk patients with acute coronary syndrome: a prospective observational study. BMJ Open. 2017 Jul 10;7(7):e014655. doi: 10.1136/bmjopen-2016-014655. PMID 28698323